CLINICAL TRIAL: NCT04692532
Title: Time Restricted Eating for Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Krista Varady, Professor of Nutrition, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-1512
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 8-hour Time restricted eating (Experimental): Ad libitum food intake from 12-8 pm every day Fasting from 8-12 pm every day (16-h fast)
  Interventions: Other: 8-hour Time restricted eating
- Calorie restriction (Experimental): 25% energy restriction every day
  Interventions: Other: Calorie restriction
- Control (No Intervention): Usual diet, Ad libitum intake, eating within >10 hours per day

INTERVENTIONS:
Other: 8-hour Time restricted eating — Ad libitum food intake from 12-8 pm every day Fasting from 8-12 pm every day (16-h fast)
  Arms: 8-hour Time restricted eating
Other: Calorie restriction — 25% energy restriction every day
  Arms: Calorie restriction

SUMMARY:
A 12-month randomized, controlled, parallel-arm trial, divided into 2 consecutive periods: (1) 6-month weight loss period; and (2) 6-month weight maintenance, will be implemented. Adults with obesity will be randomized to 1 of 3 groups: (1) 8h-TRE, ad libitum food intake from 12pm to 8 pm, fasting from 8 pm to 12 pm daily, (2) CR, 25% energy restriction every day; or 3) control, ad libitum food intake daily, eating within more than 10 hours per day.

DETAILED DESCRIPTION:
Time restricted eating (TRE) has become a popular weight loss regimen. The sudden rise in popularity of TRE is mostly likely due to is its sheer simplicity, and the fact that it does not require individuals to count calories in order to lose weight. Participants are simply asked to consume all food within a specified time frame and fast with energy free beverages for the remaining hours of the day. Evidence shows that when people with obesity limit their eating window to 6 to 8 hours per day, they naturally reduce energy intake by 350-500 calories. From a clinical standpoint, these findings are paramount. One of the main reasons for subject attrition with traditional dieting, i.e. daily calorie restriction (CR), is frustration with having to count calories every day. TRE regimens are able to side-step this requirement by allowing participants to simply "watch the clock" instead of monitoring calories, while still producing significant weight loss and metabolic health improvements. This feature of TRE has the potential to improve long-term adherence to the diet, and in turn produce lasting weight control in adults with obesity.

Accordingly, we conducted a one-year, randomized, controlled trial to compare the effects of late TRE (eating all food between 12:00 pm to 8:00 pm, without calorie counting), versus CR (25% energy restriction daily), and a control group eating over a period of 10 or more hours, on body weight and metabolic risk factors in a diverse group of American adults with obesity. We hypothesized that the TRE group would achieve greater weight loss, and experience more pronounced improvements in insulin sensitivity during the 6-month weight loss phase, compared to CR and control participants. We also hypothesized that the TRE group would better maintain their weight loss and sustain their improvements in insulin sensitivity during the 6-month weight maintenance phase, when compared to the CR and control participants.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 to 65 years old
* BMI between 30 and 50 kg/m2
* Sedentary or lightly active (<60 minutes/week of light activity for the 3 months prior to the study)

Exclusion criteria:

* • Type 1 DM or Type 2 DM
* History of eating disorders (anorexia, bulimia, or binge eating disorder)
* Are not weight stable for 3 months prior to the beginning of study (weight gain or loss > 4 kg)
* Are not able to keep a food diary or activity log for 7 consecutive days during screening
* Are taking drugs that influence study outcomes (weight loss, glucose-lowering medications)
* Are perimenopausal or have an irregular menstrual cycle (menses that does not appear every 27-32 days)
* Are eating within less than a 10-hour window at baseline
* Are pregnant, or trying to become pregnant
* Are night shift workers
* Are smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Measured at month 0, 6 and 12
  Measured by an electronic scale

SECONDARY OUTCOMES:
Change in fat mass, lean mass, visceral fat mass | Measured at month 0, 6 and 12
  Measured by DXA
Change in bone mineral density | Measured at month 0, 6 and 12
  Measured by DXA
Change in waist circumference | Measured at month 0, 6 and 12
  Measured by a measuring tape
Change in Insulin resistance | Measured at month 0, 6 and 12
  Measured by HOMA-IR
Change in Insulin sensitivity | Measured at month 0, 6 and 12
  Measured by QUICKI
Change in Fasting glucose | Measured at month 0, 6 and 12
  Measured by a commercial lab (Medstar, IL)
Change in HbA1c | Measured at month 0, 6 and 12
  Measured by a commercial lab (Medstar, IL)
Change in Fasting insulin | Measured at month 0, 6 and 12
  Measured by a commercial lab (Medstar, IL)
Change in Blood pressure | Measured at month 0, 6 and 12
  Measured by a blood pressure cuff
Change in Heart rate | Measured at month 0, 6 and 12
  Measured by a blood pressure cuff
Change in Plasma lipids (LDL cholesterol, HDL cholesterol, triglycerides) | Measured at month 0, 6 and 12
  Measured by a commercial lab (Medstar, IL)
Change in inflammatory markers (TNF-apha, IL-6, IL-10, IL-B, hs-CRP) | Measured at month 0, 6 and 12
  Measured by ELISA
Change in oxidative stress | Measured at month 0, 6 and 12
  Measured by ELISA
Change in estradiol levels (ng/ml) | Measured at month 0, 6 and 12
  Measured by ELISA
Change in testosterone levels (ng/ml) | Measured at month 0, 6 and 12
  Measured by ELISA
Change in dehydroepiandrosterone (DHEA) levels (ng/ml) | Measured at month 0, 6 and 12
  Measured by ELISA
Change in sex hormone binding globulin (SHBG) levels (ng/ml) | Measured at month 0, 6 and 12
  Measured by ELISA
Change in progesterone levels (ng/ml) | Measured at month 0, 6 and 12
  Measured by ELISA
Change in energy and nutrient intake | Measured at month 0, 6 and 12
  Measured by 7-day food record
Change in physical activity (steps/d) | Measured at month 0, 6 and 12
  Measured by pedometer
Change in the daily eating window | Measured at month 0, 6 and 12
  Measured by questionnaire (assesses the time the participant started and stopped eating each day)
Change in sleep quality | Measured at month 0, 6 and 12
  Measured by Pittsburgh Sleep Quality Index (PSQI), total score of 0-21. A PSQI total score greater than 5 indicates poor sleep quality.
Change in insomnia severity | Measured at month 0, 6 and 12
  Measured by Insomnia Severity Index (ISI), total score of 0-28. The total score for the ISI is interpreted as follows: no clinically significant insomnia (0-7), sub-threshold insomnia (8-14), moderate severity insomnia (15-21), and severe insomnia (22-28).
Change in risk of sleep apnea | Measured at month 0, 6 and 12
  Measured by Berlin Questionnaire, measures the presence or absence of sleep apnea
Change in mood | Measured at month 0, 6 and 12
  Measured by Beck Depression Inventory II (BDI-II) 25: total score 0-100. Higher scores mean worse outcome. Also measured by the Profile of Mood States (POMS)total score 0-100. Higher scores mean worse outcome.
Change in quality of life | Measured at month 0, 6 and 12
  Measured by the Short Form Survey (SF-36): total score 0-100. Higher scores mean worse outcome.
Adverse events | Measured at month 0, 6 and 12
  Measured by questionnaire
Change in appetite | Measured at month 0, 6 and 12
  Measured by Visual analog scale (VAS). Scored from 0-100. Higher score means higher appetite.
Change in eating disorder symptoms | Measured at month 0, 6 and 12
  Measured by Multifactorial Assessment of Eating Disorders Symptoms (MAEDS), total score of 0-100, Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Varady, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin S, Cienfuegos S, Ezpeleta M, Pavlou V, Runchey MC, Varady KA. Effect of time restricted eating versus daily calorie restriction on sex hormones in males and females with obesity. medRxiv [Preprint]. 2024 May 15:2024.05.15.24307415. doi: 10.1101/2024.05.15.24307415. PMID 38798539
- [Derived] Lin S, Cienfuegos S, Ezpeleta M, Gabel K, Pavlou V, Mulas A, Chakos K, McStay M, Wu J, Tussing-Humphreys L, Alexandria SJ, Sanchez J, Unterman T, Varady KA. Time-Restricted Eating Without Calorie Counting for Weight Loss in a Racially Diverse Population : A Randomized Controlled Trial. Ann Intern Med. 2023 Jul;176(7):885-895. doi: 10.7326/M23-0052. Epub 2023 Jun 27. PMID 37364268